CLINICAL TRIAL: NCT02954952
Title: EEG Data Collection to Evaluate New Patient State Index Performance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RAMS0005
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Standard of care (baseline) (Other): Subjects will receive the Sedline sensor. The anesthesiologist will be blinded to the PSI Rev 1.X score and the raw EEG data from the Masimo device. Anesthesia management will be in accordance with standard of care protocols and procedures.
  Interventions: Device: PSI Rev 1.X
- PSI Rev 1.X (Experimental): The anesthesiologist will be monitoring subjects using an old version of PSI (Rev 1.X).
  Interventions: Device: PSI Rev 1.X
- PSI Rev 2.X (Experimental): The anesthesiologist will be monitoring subjects using a new version of PSI (Rev 2.X).
  Interventions: Device: PSI Rev 2.X

INTERVENTIONS:
Device: PSI Rev 1.X — PSI Rev 1.X is an older version of the PSI measurement.
  Arms: PSI Rev 1.X; Standard of care (baseline)
Device: PSI Rev 2.X — PSI Rev 2.X is a newer version of the PSI measurement.
  Arms: PSI Rev 2.X

SUMMARY:
This is a prospective, single-center, cohort study in patients undergoing surgical procedures to collect data using Masimo SedLine EEG device in order to evaluate a newer version of PSI measurement against an older version of PSI measurement.

ELIGIBILITY:
Inclusion Criteria:

* ASA status of I, II, or III.
* Subjects undergoing general surgery.
* neurologically intact patients (e.g. no history or presence of traumatic brain injuries, neurological diseases, etc.).

Exclusion Criteria:

* subjects with any deformities, diseases, or for any other reason that may present proper fit and application of SedLine sensors.
* inability to obtain subject's physiological, vital, demographics, and real time anesthesia data.
* Subjects who are pregnant.
* known history of drug abuse.
* subjects deemed not suitable for study at the discretion of the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ramsay, M.D., Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care (Baseline) | PSI Rev 1.X | PSI Rev 2.X
Started | 36 | 5 | 3
Completed | 35 | 4 | 3
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — No data collected | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (Baseline) | PSI Rev 1.X | PSI Rev 2.X | Total
Number analyzed (Participants) | 36 | 5 | 3 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 4 | 1 | 30
  >=65 years | 11 | 1 | 2 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (14.3) | 55.2 (15.5) | 67 (2.6) | 56.5 (14.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 22 | 4 | 1 | 27
  Male | 13 | 1 | 2 | 16
  Unknown | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 27 | 5 | 3 | 35
  Black or African American | 6 | 0 | 0 | 6
  Hispanic | 2 | 0 | 0 | 2
  Unknown | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 5 | 3 | 44

OUTCOME MEASURES:

1. Primary Outcome: Wake up Times, PSI 1.X vs. PSI 2.X
Description: Compare the length of time from when the anesthesia has ended to the time of Return of Consciousness (ROC) between the PSI 1.X group and the PSI 2.X group.
Time Frame: From the end of anesthesia to the time of Return of Consciousness
Population: Data were not collected.
Arm/Group | Standard of Care (Baseline) | PSI Rev 1.X | PSI Rev 2.X
Number analyzed (Participants) | 0 | 0 | 0

2. Other Pre Specified Outcome: Total Anesthesia Drug Used, PSI 1.X vs. PSI 2.X
Description: Compare the total amount of anesthesia drug used between the PSI 1.X group and the PSI 2.X group.
Time Frame: Through study completion
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Frequency of Somatic Events, PSI 1.X vs. PSI 2.X
Description: Compare the frequency of somatic events between the PSI 1.X group and the PSI 2.X group.
Time Frame: Through study completion
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of SedLine sensor application until the sensor is removed when the subject wakes up from anesthesia.
Arm/Group | Standard of Care (Baseline) | PSI Rev 1.X | PSI Rev 2.X
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 0/36 | 0/5 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can initiate publication after 12 months of study completion or early termination (whichever is applicable). The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT02954952/Prot_SAP_000.pdf